CLINICAL TRIAL: NCT04844268
Title: Phase 1, Randomized, Double-Blind, Dose-Escalation Study to Evaluate the Safety, Reactogenicity and Immunogenicity of Nanoparticle Carrier-Formulated Self-Replicating Replicon RNA (repRNA) Vaccine in Healthy Adults
Brief Title: Study to Assess Safety, Reactogenicity and Immunogenicity of the VACCINE RNA MCTI CIMATEC HDT (HDT-301) Vaccine Against COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SENAI CIMATEC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIMATEC01
Record Dates: First submitted 2021-04-08; First posted 2021-04-14 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: SARS-CoV-2
MeSH Terms: interventions — repRNA-CoV2S vaccine; Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding was done to all cohorts. Subjects, clinical study staff, statisticians, and investigators were masked to treatment assignment. Laboratory staff that manipulates the vaccine and the placebo were not blinded.
  Subjects received injections of either vaccine or placebo, delivered in the deltoid muscle in accordance with the study protocol. In order to internal contents were not differentiated, the injections were applied with opaque syringes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Intramuscular (IM) injection of VACCINE RNA MCTI CIMATEC HDT(HDT-301) at a dose of 1 µg. Participants will be randomized (4:1 ratio for active vaccine:placebo) with equal probability of receiving a schedule of two doses, of the same concentration, on days 1 and 28 (group 1) or 1 and 56 (group 2), or a schedule of single-dose administration (group 3).
  Interventions: Biological: Cohort 1 VACCINE RNA MCTI CIMATEC HDT (HDT-301) vaccine; Biological: Placebo
- Cohort 2 (Experimental): Intramuscular (IM) injection of VACCINE RNA MCTI CIMATEC HDT(HDT-301) at a dose of 5 µg. Participants will be randomized (4:1 ratio for active vaccine:placebo) with equal probability of receiving a schedule of two doses, of the same concentration, on days 1 and 28 (group 1) or 1 and 56 (group 2), or a schedule of single-dose administration (group 3).
  Interventions: Biological: Cohort 2 RNA VACCINE MCTI CIMATEC HDT(HDT-301) vaccine; Biological: Placebo
- Cohort 3 (Experimental): Intramuscular (IM) injection of VACCINE RNA MCTI CIMATEC HDT(HDT-301) at a dose of 25 µg. Participants will be randomized (4:1 ratio for active vaccine:placebo) with equal probability of receiving a schedule of two doses, of the same concentration, on days 1 and 28 (group 1) or 1 and 56 (group 2), or a schedule of single-dose administration (group 3).
  Interventions: Biological: Cohort 3 VACCINE RNA MCTI CIMATEC HDT(HDT-301) vaccine; Biological: Placebo
- Placebo (Placebo Comparator): Intramuscular (IM) injection of saline (0.9% sodium chloride). Participants will be randomized (4:1 ratio for active vaccine:placebo) with equal probability of receiving a schedule of two doses, of the same concentration, on days 1 and 28 (group 1) or 1 and 56 (group 2), or a schedule of single-dose administration (group 3).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Cohort 1 VACCINE RNA MCTI CIMATEC HDT (HDT-301) vaccine — Intramuscular injections of 1 µg of novel Lipid-Inorganic Nanoparticle (LION) formulated replicating RNA-based vaccine (VACCINE RNA MCTI CIMATEC HDT (HDT-301)) at a dose of 1 µg on days 1 and 28 (group 1) or 1 and 56 (group 2), or a schedule of single dose administration (group 3).
  Arms: Cohort 1
Biological: Cohort 2 RNA VACCINE MCTI CIMATEC HDT(HDT-301) vaccine — Intramuscular injections of 5 µg of novel Lipid-Inorganic Nanoparticle (LION) formulated replicating RNA-based vaccine (VACCINE RNA MCTI CIMATEC HDT(HDT-301)) at a dose of 5 µg on days 1 and 28 (group 1) or 1 and 56 (group 2), or a schedule of single dose administration (group 3).
  Arms: Cohort 2
Biological: Cohort 3 VACCINE RNA MCTI CIMATEC HDT(HDT-301) vaccine — Intramuscular injections of 25 µg of novel Lipid-Inorganic Nanoparticle (LION) formulated replicating RNA-based vaccine (VACCINE RNA MCTI CIMATEC HDT(HDT-301)) at a dose of 25 µg on days 1 and 28 (group 1) or 1 and 56 (group 2), or a schedule of single dose administration (group 3).
  Arms: Cohort 3
Biological: Placebo — Intramuscular (IM) injection of saline (0.9% sodium chloride) on days 1 and 28 (group 1) or 1 and 56 (group 2), or a schedule of single dose administration (group 3), in each cohort.

SUMMARY:
This is a phase I, double-blind, placebo-controlled,dose-ranging clinical trial in healthy males and non-pregnant females, 18 to 55 years of age. The trial is designed to assess the safety, reactogenicity, and immunogenicity of VACCINE RNA MCTI CIMATEC HDT(HDT-301), which is a novel Lipid-Inorganic Nanoparticle (LION) formulated replicating RNA-based vaccine that encodes for a full-length spike (S) protein of the SARS-CoV-2 virus. As a replicating mRNA vaccine, VACCINE RNA MCTI CIMATEC HDT(HDT-301) has the potential to allow the advantages of dose sparing, and possibly administration as a single dose, compared with other mRNA platforms.

Enrollment will occur at one domestic site. A total of 90 healthy subjects will receive multiple dosages of intramuscular (IM) injections of VACCINE RNA MCTI CIMATEC HDT(HDT-301). Participants will be enrolled sequentially in three dose cohorts (cohort 1 = 1 µg, cohort 2 = 5 µg, and cohort 3 = 25 µg), with each cohort consisting of a total of 30 subjects. Within each dose cohort, participants will be randomized (4:1 ratio for active vaccine:placebo) with equal probability of receiving a schedule of two doses, of the same concentration, on days 1 and 28 (group 1) or 1 and 56 (group 2), or a schedule of single dose administration (group 3) VACCINE RNA MCTI CIMATEC HDT(HDT-301). The main objective is to evaluate the safety and reactogenicity of 3 dose vaccination schedule of VACCINE RNA MCTI CIMATEC HDT(HDT-301) and 1 dose of placebo in healthy adults.

Safety and tolerability will be the primary endpoint assessed by incidence of adverse events for each dose through 12 months after the vaccination. Scheduled interim immunogenicity evaluations will be conducted for pre-specified timepoints as secundary and exploratory endpoints.

DETAILED DESCRIPTION:
In this phase 1 dose-ranging study, 3 dosage cohorts (1 µg, 5 µg, 25 µg), 90 subjects will be randomized (4:1 ratio for active vaccine:placebo) with equal probability of receiving a two-dose schedule of the same concentration, 28 days (group 1) or 56 days (group 2 ) after the first dose, or, a single dose schedule (group 3). For each of the three cohorts, for safety reasons, 1 sentinel subject will be registered initially, and will be vaccinated with the experimental drug, and will be followed up until day 8 (seven days after the first dose). If any criterion for interruption does not occur by day 8, 4 more sentinel subjects will be recruited and included in the study.

This means that once the first sentinel subject must receive the study vaccine, of the 4 sentinel participants enrolled later, 3 will receive the vaccine and 1 will receive the placebo (0.9% sodium chloride solution). Only then, after the 7-day follow-up period of the last sentinel subject, if no stopping rule is identified, the recruitment and registration of the remaining 25 subjects will proceed.

After cohort 1 has been registered, cohort 2 will be registered in a similar manner, with the first sentinel subject being registered after a 7-day observation period followed by the vaccination of the last subject in cohort 1. Cohort 3 will be registered in a similar manner after cohort 2.

There is a placebo group in each cohort in order to compare and improve the assessment of causality of adverse events.

Double blinding was done to all cohorts. Subjects, clinical study staff, statisticians, and investigators were masked to treatment assignment. Laboratory staff that manipulates the vaccine and the placebo were not blinded.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet ALL of the following criteria to be eligible for inclusion in this phase I study.

i. Men and women ≥ 18 years to ≤ 55 years of age; ii. Must be generally healthy as confirmed by a medical history and physical examination for study entry; iii. Subjects who have not been previously immunized with any SARS-CoV-2 vaccine OR subjects who have been immunized with SARS-CoV-2 vaccine based inactivated virus technology at least 3 months from the administration of the second dose and have neutralizing antibody titers less than or equal to 40% in plasma samples tested at 1:40 dilution; iv. Women of childbearing age and of childbearing potential must present during the screening period and on the day of each vaccination the result of a pregnancy test (serum test) with a negative result, as well as not be breastfeeding; in addition, to enroll in the study as volunteers, women who have sex with men must necessarily use one of the contraceptive methods listed below at the time of enrollment and up to 60 days after the last injection of the vaccine (this 60-day interval has been defined as a safety criterion): hormonal (e.g., oral, transdermal, intravaginal, implant, or injection); double barrier (i.e., condom, diaphragm, or cervical cap with spermicide); intrauterine device (IUD) or intrauterine system (IUS); vasectomized (6 months minimum) or abstinent partner; bilateral tubal ligation (if no conception post-procedure); tubal occlusion or bilateral salpingectomy. These precautions are necessary because of unknown effects that Vaccine RNA MCTI CIMATEC HDT may cause in a fetus or newborn. Women will be considered out of the potential to become pregnant if they are postmenopausal (defined as spontaneous amenorrhea of at least 12 months and confirmed with follicle-stimulating hormone concentrations >40 mUI/ml) or have documented hysterectomy and/or oophorectomy; and, non-sterile men who agree to use adequate contraception with their partner during and up to 60 days after the last injection of the study vaccine; v. The following laboratory test values for screening must be within normal limits or not clinically significant, as determined by the Researcher and approved by the Medical Monitor: sodium, potassium, Glutamic-Oxalacetic Transaminase (GOT), Glutamic-Pyruvic Transaminase (GPT), total bilirubin, alkaline phosphatase, creatinine, fasting glucose, total WBC, hemoglobin, and platelet count. Abnormal results may be repeated once for confirmation at the discretion of the Researcher; vi. The following serological tests must be negative: HIV 1/2 antibody, hepatitis B surface antigen (HBsAg) and hepatitis C virus (HCV) antibody; vii. Negative test for recreational drugs and alcohol according to the standards of the Clinical Research Unit; viii. Normal or not clinically significant urine test as determined by the clinician or designee. Abnormal results may be repeated at the discretion of the Researcher; ix. Must present blood count within normal limits up to 10 days prior to administration of the first dose of the Vaccine RNA MCTI CIMATEC HDT; x. Must present negative RT-PCR test for SARS-CoV-2 24 to 48 h before administration of the study vaccine and absence of signs and symptoms compatible with COVID-19 (e.g. fever, cough, shortness of breath, chills, etc.); xi. Must be able to complete the Mnemonic Adverse Event Questionnaire (MMEA) (Appendix 1); xii. Must give informed consent, be able and willing to make all evaluation visits, be accessible by phone or personal contact by the local study team, and have a permanent address.

Exclusion Criteria:

Individuals who meet ANY of the following criteria below will be excluded from the study (ineligible).

i. Participation in another experimental protocol and/or receipt of any investigational product within the last 3 months prior to screening; ii. Individuals infected with SARS-CoV-2 confirmed by RT-PCR; iii. Treatment with immunosuppressive drugs (e.g., oral or injectable steroidal anti-inflammatory drugs, such as prednisone, or high-dose inhalation) or cytotoxic therapies (e.g., chemotherapeutic drugs or radiation) within the last 6 months prior to screening; iv. Individuals who have received transfusion of blood, plasma, or immunoglobulins in the last 3 months prior to screening; v. Donation of blood products (platelets, whole blood, plasma, etc.) in the last month before screening (1 month before screening); vi. Received any vaccinations in the last month before screening or have any immunizations planned during the study, with the exception of seasonal influenza vaccine, which can be given after 30 days after the second injection of the study; vii. Individuals who have been immunized with any vaccine for SARS-CoV-2 at any time who have neutralizing antibody titers greater than 40% in plasma samples tested at 1:40 dilution; viii. History of autoimmune disease or other causes of immunosuppressive states; ix. History of any other acute or chronic disease (including cardiovascular, pulmonary, neurological, hepatic, rheumatic, hematological, metabolic or renal disorders, uncontrolled hypertension) or use of medications that, in the opinion of the Principal Investigator, may interfere with the safety or immunogenicity evaluation of the vaccine; x. Skin rash, tattoos or any other dermatological condition that may adversely affect the vaccine injection site or interfere with its evaluation; xi. BMI ≥ 32; xii. Hypertension (systolic > 150 or diastolic > 95); xiii. History of significant psychiatric illness with current medication use; xiv. Known or suspected alcohol or drug abuse in the last 6 months prior to screening; xv. Chronic tobacco user (> 20 packs/year); xvi. Individuals with a history of prior anaphylaxis or severe allergic reaction to unknown vaccines or allergens; xvii. Individuals unlikely to cooperate with the requirements of the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of a schedule of 2 administrations and a schedule of one administration of VACCINE RNA MCTI CIMATEC HDT | day 1 and 28 days after the each vaccination until day 84
  Incidence of adverse event, serious adverse event, adverse event of special interest and adverse event that requires medical evaluation
Reactogenicity of a schedule of 2 administrations and a schedule of one administration of VACCINE RNA MCTI CIMATEC HDT . | Day 2 and 7 after each vaccination
  local and sistemic adverse events, laboratorial anormalities

SECONDARY OUTCOMES:
Immunogenicity of a schedule of 2 administrations and a schedule of one administration of VACCINE RNA MCTI CIMATEC HDT (IgG) | During 12 months of follow up
  Geometric means of IgG titers by ELISA to the SARS-CoV-2 Spike (S) protein at multiple time points
Immunogenicity of a schedule of 2 administrations and a schedule of one administration of VACCINE RNA MCTI CIMATEC HDT (neutralizing antibodies) | During 12 months of follow up
  Geometric means of specific neutralizing antibodies titers to the SARS-CoV-2 at multiple time points
mmunogenicity of a schedule of 2 administrations and a schedule of one administration of VACCINE RNA MCTI CIMATEC HDT : proportion of IgG antibodies titers | Day 1 (cohort 1, 2 and 3), day 29 (cohort 1), day 57 (cohort 2) and 28 days after the second vaccination ( cohort 1: day 57 and cohort 2: day 85)
  Proportion of subjects with a ≥4-fold increase in IgG antibody titer to SARS-CoV-2 by ELISA
Immunogenicity of a schedule of 2 administrations and a schedule of one administration of VACCINE RNA MCTI CIMATEC HDT: proportion of specific neutralizing antibodies titers | Day 1 (cohort 1, 2 and 3), day 29 (cohort 1), day 57 (cohort 2) and 28 days after the second vaccination ( cohort 1: day 57 and cohort 2: day 85)
  Proportion of subjects with a ≥4-fold increase in specific neutralizing antibodies titers to SARS-CoV-2 by ELISA

OTHER OUTCOMES:
Immunogenicity of a schedule of 2 administrations and a schedule of one administration of VACCINE RNA MCTI CIMATEC HDT (IgM, IgA and IgG subtipes) | During 12 months of follow up
  Geometric means of IgM, IgA and IgG subtipes (IgG1, IgG2, IgG3 e IgG4) titers by ELISA specific to the SARS-CoV-2 at multiple time points
Immunogenicity of a schedule of 2 administrations and a schedule of one administration of VACCINE RNA MCTI CIMATEC HDT (IgM, IgA and IgG subtipes): proportion | Day 1, 8,29,57,85,114, 180 and 365 for all cohorts. Day 36 for cohort 1 and 64 for cohort 2
  Proportion of subjects with a ≥4-fold increase in IgM, IgA and IgG subtipes (IgG1, IgG2, IgG3 e IgG4) titers specific for SARS-CoV-2 by ELISA
Immunogenicity of a schedule of 2 administrations and a schedule of one administration of VACCINE RNA MCTI CIMATEC HDT : T cells response | Day 1, 8,29,57,85,114, 180 and 365 for all cohorts. Day 36 for cohort 1 and 64 for cohort 2
  Levels of Interferon Gamma, Interleukins 2, 5 and 13, tumor necrosis factor, CD3, CD4 and CD8

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Badaró, PhD, Principal Investigator — Principal Investigator; Steven Reed, PhD, Study Chair — Study collaborator
Locations (1):
- Hospital da Bahia, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No